CLINICAL TRIAL: NCT04499196
Title: Prospective Study of Glucocorticoids as a Mechanism to Treat Pulmonary Hypertension
Brief Title: Glucocorticoids and Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: LD2020
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Hypertension Due to Lung Diseases and Hypoxia; Pulmonary Hypertension; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Hypoxia; Hypertension, Pulmonary; Bronchopulmonary Dysplasia | interventions — Glucocorticoids

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: GlucoCorticoid — Administering glucocorticoid

SUMMARY:
Pediatric idiopathic pulmonary hypertension has significant morbidity and mortality. An ever expanding body of knowledge indicates the important contribution of inflammation to pathogenesis and successful treatment with glucocorticoids. Over the last several years the investigators have utilized steroids in patients with severe pulmonary hypertension as part of a treatment regimen. These basic science studies possibly identifies a biochemical etiology for the development of disease and may also be impacted by the administration of steroids. Additionally, there is a commercially available assay which tests for all of the above molecules.

ELIGIBILITY:
Inclusion Criteria:

* premature, BPD, >36 wga
* pulmonary hypertension evidence by echocardiogram

Exclusion Criteria:

* poor ventilation/oxygenation

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates with BPD
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-07-29 (Estimated); Study Completion 2022-07-29 (Estimated)

PRIMARY OUTCOMES:
Echo estimation of RV pressure | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuder RM, Groves B, Badesch DB, Voelkel NF. Exuberant endothelial cell growth and elements of inflammation are present in plexiform lesions of pulmonary hypertension. Am J Pathol. 1994 Feb;144(2):275-85. PMID 7508683
- [Background] Perros F, Dorfmuller P, Montani D, Hammad H, Waelput W, Girerd B, Raymond N, Mercier O, Mussot S, Cohen-Kaminsky S, Humbert M, Lambrecht BN. Pulmonary lymphoid neogenesis in idiopathic pulmonary arterial hypertension. Am J Respir Crit Care Med. 2012 Feb 1;185(3):311-21. doi: 10.1164/rccm.201105-0927OC. Epub 2011 Nov 22. PMID 22108206
- [Background] Savai R, Pullamsetti SS, Kolbe J, Bieniek E, Voswinckel R, Fink L, Scheed A, Ritter C, Dahal BK, Vater A, Klussmann S, Ghofrani HA, Weissmann N, Klepetko W, Banat GA, Seeger W, Grimminger F, Schermuly RT. Immune and inflammatory cell involvement in the pathology of idiopathic pulmonary arterial hypertension. Am J Respir Crit Care Med. 2012 Nov 1;186(9):897-908. doi: 10.1164/rccm.201202-0335OC. Epub 2012 Sep 6. PMID 22955318
- [Background] Stenmark KR, Meyrick B, Galie N, Mooi WJ, McMurtry IF. Animal models of pulmonary arterial hypertension: the hope for etiological discovery and pharmacological cure. Am J Physiol Lung Cell Mol Physiol. 2009 Dec;297(6):L1013-32. doi: 10.1152/ajplung.00217.2009. Epub 2009 Sep 11. PMID 19748998
- [Background] Langleben D, Reid LM. Effect of methylprednisolone on monocrotaline-induced pulmonary vascular disease and right ventricular hypertrophy. Lab Invest. 1985 Mar;52(3):298-303. PMID 3156262
- [Background] Wang W, Wang YL, Chen XY, Li YT, Hao W, Jin YP, Han B. Dexamethasone attenuates development of monocrotaline-induced pulmonary arterial hypertension. Mol Biol Rep. 2011 Jun;38(5):3277-84. doi: 10.1007/s11033-010-0390-x. Epub 2011 Mar 23. PMID 21431360
- [Background] Ogawa A, Nakamura K, Mizoguchi H, Fujii N, Fujio H, Kusano KF, Ohe T, Ito H. Prednisolone ameliorates idiopathic pulmonary arterial hypertension. Am J Respir Crit Care Med. 2011 Jan 1;183(1):139-40. doi: 10.1164/ajrccm.183.1.139. No abstract available. PMID 21193794
- [Background] Ogawa A, Nakamura K, Matsubara H, Fujio H, Ikeda T, Kobayashi K, Miyazaki I, Asanuma M, Miyaji K, Miura D, Kusano KF, Date H, Ohe T. Prednisolone inhibits proliferation of cultured pulmonary artery smooth muscle cells of patients with idiopathic pulmonary arterial hypertension. Circulation. 2005 Sep 20;112(12):1806-12. doi: 10.1161/CIRCULATIONAHA.105.536169. Epub 2005 Sep 12. PMID 16157769
- [Background] Aggarwal M, Grady RM. Glucocorticoids for treating paediatric pulmonary hypertension: a novel use for a common medication. Cardiol Young. 2017 Sep;27(7):1410-1412. doi: 10.1017/S1047951117000464. Epub 2017 May 16. PMID 28506331